CLINICAL TRIAL: NCT02075359
Title: Novel Models to Predict Energy Expenditure and Physical Activity in Preschoolers
Brief Title: Energy Expenditure and Physical Activity in Preschoolers
Acronym: LILCAL
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Drexel University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nancy Butte, Principal investigator and Professor, Baylor College of Medicine
Other Study IDs: H12067; R01DK085163 (NIH)
Record Dates: First submitted 2014-02-21; First posted 2014-03-03 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Total Energy Expenditure; Physical Activity Levels; Body Mass Index; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preschoolers: Preschoolers, ages 3 to 5

SUMMARY:
The purpose of this study is to calibrate the Actigraph, Respironics and CamNtech monitors, in a wide range of children using energy expenditure measured by respiration calorimetry. Energy expenditure will be predicted from the combination of heart rate and activity measured by accelerometry. Prediction equations for energy expenditure will be tested and validated against a stable isotope method called doubly labeled water for the measurement of free-living total energy expenditure.

DETAILED DESCRIPTION:
In this study, the investigators will apply advanced technology (fast-response room calorimetry, doubly labeled water (DLW), accelerometers and miniaturized HR monitors) and sophisticated mathematical modeling techniques (cross-sectional time series, CSTS and multivariate adaptive regression splines, MARS) to develop and validate prediction models that capture the dynamic nature of physical activity (PA) and energy expenditure (EE) in preschool-aged children. CSTS and MARS models for the assessment of PA based on activity energy expenditure (AEE) and for the prediction of minute-by-minute EE will be developed in 100 preschool-aged children using 12-h room respiration calorimetry as the criterion method and validated in an independent sample (n=50) against 12-h room respiration calorimetry and the 7-d DLW method. In addition, the investigators will develop algorithms for the classification of PA levels and sleep/awake periods using statistical and machine learning methods and incorporate the results into our prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between the ages of 3-5 years will be recruited from the local community. A total of 150 children will be studied. In Phase I, 100 children will be studied and in Phase II 50 children will be studied.

Exclusion Criteria:

* any medical illness or medication affecting growth or limiting participation in physical activities or sports.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Child (3-5 years)
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | up to 1 year
  Energy expenditure will be measured by calorimetry and the doubly labeled water method.

SECONDARY OUTCOMES:
physical activity | Up to 1 year
  The physical activity level of children will be measured by accelerometry and heart rate monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Butte, Ph.D, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States